CLINICAL TRIAL: NCT06176456
Title: Interventional Triple-negative Placebo-controlled Personalized Prospective Study "Evaluation of the Efficacy and Safety of Noninvasive Neuromodulation of TMS in Subjects With Catatonia"
Brief Title: Personalized Prospective Study Evaluation of the Efficacy and Safety of Noninvasive Neuromodulation of TMS in Subjects With Catatonia
Acronym: RECATA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow Psychiatric Hospital No. 1 Named after N.A. Alexeev (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RECATA
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Catatonia; Schizophrenia; Schizo Affective Disorder; Bipolar Affective Disorder
MeSH Terms: conditions — Catatonia; Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: The design of the study involves following stages:
  * diagnostic stage and randomization;
  * 10 sessions of placebo-controlled stimulation protocols (high- and low-frequency magnetic pulses)
  * primary analysis of the effectiveness of protocols after 10 sessions of stimulation, followed by the transfer of all patients, including the placebo group to the most effective stimulation regiment (20 sessions of active neuromodulation)
  * final analysis of the effectiveness after 20 sessions of TMS and follow-up period (visits after 1 month and 6 months)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 sessions with a frequency of 1 Hz (Active Comparator): 10 sessions with a frequency of 1 Hz with an amplitude of 120% of the evoked motor response in the projection of the left Dorsolateral prefrontal cortex 1600 pulses per session with total duration of procedure ~ 20 minutes
  Interventions: Diagnostic Test: rTMS
- 10 sessions with a frequency of 20 Hz (Active Comparator): 10 sessions with a frequency of 20 Hz with an amplitude of 120% of the evoked motor response in the projection of Dorsolateral prefrontal cortex (1600 pulses per session with total duration of the procedure ~ 20 minutes)
  Interventions: Diagnostic Test: rTMS
- 10 placebo sessions (Placebo Comparator): The coil emits sound and tactile artifacts indistinguishable from therapeutic ones, but without a magnetic pulses.
  Interventions: Other: Placebo

INTERVENTIONS:
Diagnostic Test: rTMS — Active regiment
  Arms: 10 sessions with a frequency of 1 Hz; 10 sessions with a frequency of 20 Hz
Other: Placebo — Tactile artefacts without magnetic pulses
  Arms: 10 placebo sessions

SUMMARY:
Evaluation effectiveness and safety of TMS in subjects with catatonia

DETAILED DESCRIPTION:
Non-pharmacological strategies for influencing brain structures show great potential, particularly transcranial magnetic stimulation (TMS), which allows targeting specific areas of the brain and activating neuroplastic processes that contribute to the restoration of lost functions. According to study hypothesis, therapy for catatonia is possible through the stimulation of the dorsolateral prefrontal cortex (DLPFC), given its accessibility and role in the syndrome's development because. It has been established that a key process in the pathogenesis of catatonia is the disruption of the structural-functional connectivity and activity of several regions within the fronto-temporal network

The design of the study involves following stages:

* diagnostic stage and randomization
* two personalized stimulation protocols (high- and low-frequency delivery of magnetic pulses) with placebo control
* initial analysis of the effectiveness of protocols after 10 sessions of stimulation, followed by the transfer of all patients, including the placebo group to the most effective protocol.
* the stage of active neuromodulation of 20 sessions (4 weeks) according to the protocol of effective stimulation regiment
* final analysis of the effectiveness after 20 sessions of TMS, as well as after 1 and 6 months

ELIGIBILITY:
Inclusion Criteria:

Verified diagnosis of schizophrenic or affective spectrum (schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder)

Patient's ability (possibly accompanied by caregivers) to undergo diagnostic and therapeutic procedures;

The presence of residual catatonia in the form of such psychomotor anomalies as:

* disorganisation of thinking with speech disturbance with verbigerations and/or sperrungs
* hypo- and hyperkinetic psychomotor phenomena;
* substupor without disturbance of consciousness;
* elective mutism;
* echo phenomena (echolalia and/or echopraxia);
* phenomena of "wax flexibility"
* speech and behavioral stereotypy
* pathetic exaltation phenomena
* the phenomenon of irritative asthenia
* dysuric phenomena (monotonous activity and rigidity of affect)

Exclusion Criteria:

* patient's refusal to participate in the study
* acute hallucinatory-delusional symptoms
* suicide risk
* a patient taking prohibited therapy products
* neuroleptic complications of antipsychotic therapy
* irritative asthenia
* dysuric phenomena by the type of monotonous activity and rigidity of affect

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The rate of onset of the primary response | 6 months
  Reduction of points on the BPRS and NCRS scales to 70% of the initial
The number of patients with a positive effect of therapy | 6 months
  Reduction of the total score on BFCRS and NCRS by at least 50%
The number of patient with the improvement | 6 months
  The total score for BFCRS and NCRS is no more than 3 points

CONTACTS AND LOCATIONS:
Locations (1):
- "Mental-health Clinic No.1 named N.A.Alexeev of Moscow Health Department" Moscow, Russia, Moscow, Russia

REFERENCES:
- [Background] Il'ina NA, Zakharova NV. [Long-term dyskinetic remissions in shift-like schizophrenia]. Zh Nevrol Psikhiatr Im S S Korsakova. 2010;110(12):17-23. Russian. PMID 21311482
- [Background] Solmi M, Pigato GG, Roiter B, Guaglianone A, Martini L, Fornaro M, Monaco F, Carvalho AF, Stubbs B, Veronese N, Correll CU. Prevalence of Catatonia and Its Moderators in Clinical Samples: Results from a Meta-analysis and Meta-regression Analysis. Schizophr Bull. 2018 Aug 20;44(5):1133-1150. doi: 10.1093/schbul/sbx157. PMID 29140521
- [Background] Oulis P, Lykouras L. Prevalence and diagnostic correlates of DSM-IV catatonic features among psychiatric inpatients. J Nerv Ment Dis. 1996 Jun;184(6):378-9. doi: 10.1097/00005053-199606000-00010. No abstract available. PMID 8642390
- [Background] Aandi Subramaniyam B, Muliyala KP, Suchandra HH, Reddi VSK. Diagnosing catatonia and its dimensions: Cluster analysis and factor solution using the Bush Francis Catatonia Rating Scale (BFCRS). Asian J Psychiatr. 2020 Aug;52:102002. doi: 10.1016/j.ajp.2020.102002. Epub 2020 Apr 10. PMID 32506001
- [Background] Fink M, Taylor MA. Catatonia: subtype or syndrome in DSM? Am J Psychiatry. 2006 Nov;163(11):1875-6. doi: 10.1176/ajp.2006.163.11.1875. No abstract available. PMID 17074935
- [Background] Pommepuy N, Januel D. [Catatonia: resurgence of a concept. A review of the international literature]. Encephale. 2002 Nov-Dec;28(6 Pt 1):481-92. French. PMID 12506260
- [Background] Hirjak D, Rashidi M, Kubera KM, Northoff G, Fritze S, Schmitgen MM, Sambataro F, Calhoun VD, Wolf RC. Multimodal Magnetic Resonance Imaging Data Fusion Reveals Distinct Patterns of Abnormal Brain Structure and Function in Catatonia. Schizophr Bull. 2020 Jan 4;46(1):202-210. doi: 10.1093/schbul/sbz042. PMID 31174212
- [Background] Gansler DA, McLaughlin NC, Iguchi L, Jerram M, Moore DW, Bhadelia R, Fulwiler C. A multivariate approach to aggression and the orbital frontal cortex in psychiatric patients. Psychiatry Res. 2009 Mar 31;171(3):145-54. doi: 10.1016/j.pscychresns.2008.03.007. Epub 2009 Feb 11. PMID 19216060
- [Background] Northoff G, Kotter R, Baumgart F, Danos P, Boeker H, Kaulisch T, Schlagenhauf F, Walter H, Heinzel A, Witzel T, Bogerts B. Orbitofrontal cortical dysfunction in akinetic catatonia: a functional magnetic resonance imaging study during negative emotional stimulation. Schizophr Bull. 2004;30(2):405-27. doi: 10.1093/oxfordjournals.schbul.a007088. PMID 15279056
- [Background] Structure and Functions of the Human Prefrontal Cortex. Proceedings of a conference. New York City, New York, USA. March 2-4, 1995. Ann N Y Acad Sci. 1995 Dec 15;769:1-411. No abstract available. PMID 9729206
- [Background] Rolls ET. The orbitofrontal cortex. Philos Trans R Soc Lond B Biol Sci. 1996 Oct 29;351(1346):1433-43; discussion 1443-4. doi: 10.1098/rstb.1996.0128. PMID 8941955
- [Background] Stip E, Blain-Juste ME, Farmer O, Fournier-Gosselin MP, Lesperance P. Catatonia with schizophrenia: From ECT to rTMS. Encephale. 2018 Apr;44(2):183-187. doi: 10.1016/j.encep.2017.09.008. Epub 2017 Dec 11. PMID 29241672
- [Background] Hansbauer M, Wagner E, Strube W, Roh A, Padberg F, Keeser D, Falkai P, Hasan A. rTMS and tDCS for the treatment of catatonia: A systematic review. Schizophr Res. 2020 Aug;222:73-78. doi: 10.1016/j.schres.2020.05.028. Epub 2020 Jun 26. PMID 32600779
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Sharma A, Choudhury S, Anand N, Grover S, Singh SM. The use of rTMS in an adolescent presenting with acute catatonia: A case report. Asian J Psychiatr. 2018 Oct;37:1-2. doi: 10.1016/j.ajp.2018.07.017. Epub 2018 Aug 2. No abstract available. PMID 30086466
- [Background] Grisaru N, Chudakov B, Yaroslavsky Y, Belmaker RH. Catatonia treated with transcranial magnetic stimulation. Am J Psychiatry. 1998 Nov;155(11):1630. No abstract available. PMID 9812138
- [Background] Saba G, Rocamora JF, Kalalou K, Benadhira R, Plaze M, Aubriot-Delmas B, Januel D. Catatonia and transcranial magnetic stimulation. Am J Psychiatry. 2002 Oct;159(10):1794. doi: 10.1176/appi.ajp.159.10.1794. No abstract available. PMID 12359696
- [Background] Di Michele V, Bolino F. A novel treatment option of bipolar depression with psychotic and catatonic features. Gen Hosp Psychiatry. 2006 Jul-Aug;28(4):364-5. doi: 10.1016/j.genhosppsych.2006.05.003. No abstract available. PMID 16814640
- [Background] Kate MP, Raju D, Vishwanathan V, Khan FR, Nair, Thomas SV. Successful treatment of refractory organic catatonic disorder with repetitive transcranial magnetic stimulation (rTMS) therapy. J Neuropsychiatry Clin Neurosci. 2011 Summer;23(3):E2-3. doi: 10.1176/jnp.23.3.jnpe2. No abstract available. PMID 21948910
- [Background] Trojak B, Meille V, Bonin B, Chauvet-Geliner JC. Repetitive transcranial magnetic stimulation for the treatment of catatonia: an alternative treatment to electroconvulsive therapy? J Neuropsychiatry Clin Neurosci. 2014 Apr 1;26(2):E42-3. doi: 10.1176/appi.neuropsych.13050102. No abstract available. PMID 24763790
- [Background] Takamiya A, Kishimoto T, Watanabe K, Mimura M, Kito S. Transcranial Magnetic Stimulation for Bipolar Disorder with Catatonic Stupor: A Case Report. Brain Stimul. 2015 Nov-Dec;8(6):1236-7. doi: 10.1016/j.brs.2015.09.004. Epub 2015 Sep 7. No abstract available. PMID 26428351
- [Background] Stip E, Lesperance P, Farmer O, Fournier-Gosselin MP. First clinical use of epidural stimulation in catatonia. Brain Stimul. 2017 Jul-Aug;10(4):859-861. doi: 10.1016/j.brs.2017.03.006. Epub 2017 Apr 4. No abstract available. PMID 28462882